CLINICAL TRIAL: NCT00000202
Title: Buprenorphine Maintenance for Opioid Addicts
Brief Title: Buprenorphine Maintenance for Opioid Addicts - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-05626-1; R01DA005626 (NIH); R01-05626-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Opioid-Related Disorders
Keywords: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to evaluate the efficacy of buprenorphine and desipramine in treatment of opiate and cocaine dependence.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1988-08; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Kosten, M.D., Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, New Haven, Connecticut, United States

REFERENCES:
- [Background] J Nerv Mental Dis, 1993, 181(6) pp. 358-364; NIDA Res Mono 1993, 132:100 ; Am J Psychiatary 1993, 150:1755; Am J Addictions 1994, 3: 43-48; NIDA Res Mono 1994, 141:79; NIDA Res Mono 1995, in press.